CLINICAL TRIAL: NCT03027882
Title: Determining the Reliability and Validity of the Swing Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, AJ Lievre, Assistant Professor, Shenandoah University
Other Study IDs: ShenandoahU(3)
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Clinical Assessment
Keywords: Reliability; Validity; Functional Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

INTERVENTIONS:
Other: No Intervention — This is a reliability/validity study of a functional clinical test. There is no intervention

SUMMARY:
The purpose of this study is to examine the inter/intra rater reliability as well as the validity of the Swing Test in asymptomatic adults . In addition, this study will examine if there are musculoskeletal predictors to the movement quality of the swing test.

The Swing Test is a movement test used by physical therapists to identify movement problems during a simulated running stride

DETAILED DESCRIPTION:
Upon arrival the subject will be given a questionnaire that will collect demographic information and determine whether they meet the inclusion/exclusion criteria for the study. If the subjects meet the inclusion/exclusion criteria for the study, they will be given an informed consent form for participation and photography.

Prior to performing the swing test reflective markers will be placed on specific anatomical landmarks of the subject.

An investigator will demonstrate how to perform the Swing test. The subject will then be instructed to step onto a six inch box and asked to swing one leg forwards and backwards mimicking their running stride. After ten practice repetitions, ten repetitions will be recorded by the Vicon Motion Analysis System and 2 video cameras capturing different views. The subject will then step off the box and the reflective markers will be removed.

After the swing test, the subject will undergo a series of common musculoskeletal examination tests. The following examination tests will be performed in a random order.

The first musculoskeletal examination test is hip extension range of motion (ROM) that will be measured using a goniometer. The subject will lie on their stomach and the investigator will take the subjects hip into extension and measure their full motion.

The second examination tests is the Thomas test to determine the muscle length for rectus femoris muscle and iliotibial band. The subject will be instructed to sit on the edge of the bed and lower to supine while bringing one knee to chest. The investigator will assess the subject's lower extremity position to determine the length of the rectus femoris muscle and the iliotibial band.

The third examination test is hip strength measurements of internal rotation, external rotation, and abduction which will be measured using a handheld dynamometer. The subject will be placed on their back and their hip strength will be measured using the dynamometer. The subject will then be placed on their side where further hip strength will be assessed.

The fourth examination tests is the navicular drop test. In a seated position, a mark will be placed on the patient's navicular tubercle, which is a landmark on the inside of the foot. An index card will be placed next to the middle of the subjects foot and the height of the navicular will be marked on that index card. The subject will be instructed to stand up and the navicular height will be marked again on the index card. The difference in height between sitting and standing will be calculated.

The fifth examination test is the sorensen test to determine the endurance of the back muscles. The subject will be instructed to lie prone with their trunk off the treatment table. The subject will have arms crossed at chest, and will be instructed to maintain upper body horizontal the floor. Time will be recorded during the test and the tests will stop when the subject cannot maintain horizontal or 240 seconds is reached.

Three to five licensed physical therapists of varying levels of experience will be asked to watch the video recordings of the subject performing the swing test and rate their performance using a scoring system. Therapists who will be rating the Swing test will not have access to any data other than the videos.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older who run at least five (5) miles a week.

Exclusion Criteria:

* Subjects will be pain-free with no history of lower extremity, lumbar spine or pelvis musculoskeletal or neurological injuries in the last 6 months. Subjects will also not have a history of lumbar or lower extremity surgery in the last 6 months. Lastly, subjects will not have a history of balance impairments due to a vestibular or neurological disorder in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomatic adults over 18 who run at least 5 miles a week
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Swing Test | 10-15 minutes
  The subject will then be instructed to step onto a six inch box and asked to swing one leg forwards and backwards mimicking their running stride. After ten practice repetitions, ten repetitions will be recorded by the Vicon Motion Analysis System and 2 video cameras capturing different views. Three to five licensed physical therapists of varying levels of experience will be asked to watch the video recordings of the subject performing the swing test and rate their performance using a newly developed scoring system.

SECONDARY OUTCOMES:
Hip extension ROM | 5 minutes
  The subject will lie on their stomach and the investigator will take the subjects hip into extension and measure their full motion.
Thomas Test | 5 minutes
  To determine the muscle length for rectus femoris muscle and iliotibial band., the subject will be instructed to sit on the edge of the bed and lower to supine while bringing one knee to chest. The investigator will assess the subject's lower extremity position to determine the length of the rectus femoris muscle and the iliotibial band.
Hip strength | 5 minutes
  Hip internal rotation, external rotation, and abduction will be measured using a handheld dynamometer.
Navicular drop | 5 minutes
  In a seated position, a mark will be placed on the subjects navicular tubercle. An index card will be placed next to the middle of the subjects foot and the height of the navicular will be marked on that index card. The subject will be instructed to stand up and the navicular height will be marked again on the index card. The difference in height between sitting and standing will be calculated.
Sorensen Test | 5 minutes
  To determine the endurance of the back muscles, the subject will be instructed to lie prone with their trunk off the treatment table. The subject will have arms crossed at chest, and will be instructed to maintain upper body horizontal the floor. Time will be recorded during the test and the tests will stop when the subject cannot maintain horizontal or 240 seconds is reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenandoah University, Winchester, Virginia, United States